CLINICAL TRIAL: NCT01536626
Title: SWITCH Mixtard® 30 NovoLet® to NovoMix® 30 FlexPen®. An Observational Study
Brief Title: Switch From Premixed Human Insulin to Biphasic Insulin Aspart in the Netherlands
Acronym: SWITCH
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: BIASP-1925
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BIAsp 30 users
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Prescription at the discretion of the treating physician

SUMMARY:
This study is conducted in Europe. The aim of this observational study is to observe and investigate the process of switching from premixed human insulin 30/70 (BHI 30) to biphasic insulin aspart 30/70 (BIAsp 30) in an outpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic subjects treated with BHI 30

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with type 2 diabetes treated with BHI 30 who have been by the physician for some reason switched to BIAsp 30
Sampling Method: Non-Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2006-06-09 (Actual); Primary Completion 2007-04-10 (Actual); Study Completion 2007-04-10 (Actual)

PRIMARY OUTCOMES:
HbA1c (glycosylated haemoglobin)

SECONDARY OUTCOMES:
Number of hypoglycaemic events
Treatment satisfaction: ITSQ (Insulin Treatment Satisfaction Questionnaire)
Quality of Life (QoL) using the World Health Organization Wellbeing Index (WHO-5)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Alphen aan den Rijn, Netherlands

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com